CLINICAL TRIAL: NCT03345992
Title: A Double-Blind, Randomized, Placebo-Controlled Clinical Study of the Efficacy of Intravenous Clarithromycin as Adjunctive Treatment in Patients With Sepsis and Respiratory and Multiple Organ Dysfunction Syndrome
Brief Title: Benefit of Clarithromycin in Patients With Severe Infections Through Modulation of the Immune System
Acronym: INCLASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCLASS
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Sepsis; Pneumonia; Gram-Negative Bacteria Infection; Multiple Organ Failure; Respiratory Distress Syndrome; Mortality; Biomarkers
Keywords: Macrolides
MeSH Terms: conditions — Sepsis; Pneumonia; Gram-Negative Bacterial Infections; Multiple Organ Failure; Respiratory Distress Syndrome | interventions — Clarithromycin; Water; Injections

STUDY DESIGN:
Intervention Model Description: Patients assigned to either intravenous clarithromycin or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): After enrollment, the placebo arm will receive water for injection at a volume of 20ml diluted to a final volume of 250 ml dextrose in water 5%, infused once daily through intravenous route, within 1 hour, for a duration of four consecutive days.
  Interventions: Drug: Water for injection
- Clarithromycin (Active Comparator): After enrollment, the active drug arm will receive 1g of clarithromycin (500 mg powder for concentrate for solution for infusion per vial), dissolved into 20 ml water for injection and then diluted to a final volume of 250 ml dextrose in water 5%. This will be infused through intravenous route, once daily within 1 hour, for a duration of four consecutive days.
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Clarithromycin two vials of lyophilised powder for reconstitution as solution for IV administration per patient, once daily, for four consecutive days.
  Other Names: Klaricid; Biclar
  Arms: Clarithromycin
Drug: Water for injection — Water for injection 20 ml will be administered, diluted in D/W 5%, IV, once daily for four consecutive days
  Other Names: Sterile Water For Injection
  Arms: Placebo

SUMMARY:
High mortality associated with sepsis and Multiple Organ Dysfunction Syndrome (MODS) calls for alternative, individualized therapies in selected patients that might benefit form specific interventions. Role of macrolides as potential immunomodulatory treatment in sepsis is promising, but unclear. Subgroup analysis of previous large-scale clinical trials on patients with ventilator-associated pneumonia or gram-negative sepsis, showed that addition of clarithromycin to standard antibiotic therapy conferred a significant survival benefit in the subgroup of patients with respiratory dysfunction and MODS. The INCLASS study is aiming to assess the efficacy of intravenous treatment of clarithromycin in the reduction of 28-day mortality among patients suffering from these entities.

DETAILED DESCRIPTION:
Sepsis is a condition with actually rising incidence, estimated around 19 cases per 1000 hospitalizations per year in academic hospitals in USA and similar trends in Europe. It is associated with unacceptably high early (in-hospital) mortality of 40- 50%. Current guidelines promote best practice by early recognition and management with timely antibiotic administration, fluids, vasopressors and early identification/ control of infection source. However, in spite of adherence to more intensive and costly protocols of early goal-directed therapy, no further decrease in mortality is achieved. Syndromic approaches on sepsis and therapies targeting immune modulation are under evaluation and failures may partly be due to incomplete understanding of underlying pathophysiological mechanisms and immunological phases (pro and anti-inflammatory) of sepsis.

Macrolides, such as clarithromycin or azithromycin have been shown beneficial in reducing Chronic Obstructive Pulmonary Disease exacerbations (OR 0.55; 95% Confidence Intervals [CI] 0.39-0.77; p<0.001) partly through anti-inflammatory properties. Besides, when added to a beta-lactam regimen in community-acquired pneumonia, macrolide therapy was associated with reduced mortality risk (OR 0.67; 95% CI 0.61-0.73; p<0.001) in a recent meta- analysis of observational studies including 42942 patients. An immunomodulatory effect of macrolides, beyond their antimicrobial action may explain these findings.

Clarithromycin as adjunctive treatment to standard antibiotic therapy has been used by our group in two previous large-scale multi-center Randomised Controlled Trials (RCTs) conducted in Greece after approval from the Greek regulatory authorities. The first RCT studied 200 patients with sepsis due to Ventilator Associated Pneumonia (VAP) ( www.clinicaltrials.gov NCT00297674). Identified pathogens mainly included gram- negative bacteria i.e. Acinetobacter baumannii and Pseudomonas aeruginosa that do not belong to the usual antimicrobial spectrum of macrolides. Although 28-day mortality in both arms was similar, patients assigned to the clarithromycin arm experienced earlier weaning from mechanical ventilation and more rapid resolution of VAP, compared to the placebo arm. In the subgroup of patients with septic shock and multiple organ dysfunction syndrome (MODS), probability of sepsis-related death was significantly lower (OR 3.78 vs 19; p = 0.043). Serious adverse events (SAEs) occurred in 3 (3%) clarithromycin-treated patients, with no clear causative link with the study drug in 2 out of 3 cases. Furthermore, hospitalization costs associated clarithromycin use were significantly reduced (by 7000 euros/ patient) compared to the placebo arm.

The second multi-center RCT compared the efficacy of clarithromycin versus placebo added to standard antibiotic therapy in patients with gram-negative sepsis caused by acute pyelonephritis, intra-abdominal infections and primary gram- negative bacteremia; 600 patients were included (www.clinicaltrials.gov NCT01223690). Overall mortality at 28 days in both arms did not differ, but probability of death due to septic shock and MODS was shown once more lower in the clarithromycin-treated group (OR 3.58 vs 6.21; p = 0.036). Interestingly, survival benefit from clarithromycin was even greater in those patients suffering from adult respiratory distress syndrome (ARDS). SAEs were described in 2 (0.7%) patients treated with clarithromycin, while its use was associated with saving of a median of 1000 euros/ hospitalized patient.

Immunomodulatory effects of clarithromycin in sepsis are not yet elucidated. The analysis of circulating monocytes and of circulating cytokines of patients participating in the first RCT showed that treatment with clarithromycin was associated with a decline in Interleukin-10 (IL-10)/ Tumor Necrosis Factor-α (TNF-α) ratio, greater apoptosis of monocytes, enhanced antigen presentation capacity of monocytes, as well as improved capacity of monocytes for cytokine production suggesting an effect consistent with reversal of sepsis-induced immunosuppression. These findings in conjunction with evidence generated from in vitro and animal experiments suggest modulation of the immune response as the mechanism of action of clarithromycin.

In both RCTs, clarithromycin was administered intravenously at a dose of 1g as continuous one-hour intravenous infusion for three or four days. The drug was safe, well tolerated and cost-effective. However, benefit from treatment in both RCTs was shown only after sub-group analysis of the sub-group of patients with respiratory dysfunction and not when analysis comprised the entire study population. As a consequence, in order to consolidate the benefit of clarithromycin among patients with sepsis and respiratory dysfunction, the INCLASS study is a RCT designed to target a patient population with sepsis and respiratory dysfunction. It also targets a population with infections likely to be caused by Gram-negative bacteria that do not belong to the antimicrobial spectrum of clarithromycin. The study's aims are to assess the effect on mortality associated with the use of clarithromycin as adjunctive treatment in the above setting, as well as to provide insight on different biomarkers modification during treatment, to propose a mechanism of action of this treatment and to perform a cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Patients of both genders
* Informed consent form signed by patient or by first-degree relative in case of patient unable to consent
* Negative (blood or urinary) pregnancy test for female patients of reproductive age
* Willingness to receive contraception during and seven days after the administration of the study drug.
* Presence of one or more of the following infections: hospital-acquired pneumonia (HAP), health-care associated pneumonia (HCAP), ventilator-associated pneumonia (VAP), primary Gram-negative bacteremia and intra-abdominal infections.
* Presence of sepsis as defined by: Sequential Organ Failure Assessment (SOFA) score of 2 or more points for patients who are admitted with infection at the emergency department or increase of admission SOFA score by 2 or more points consequent to infection, for patients already hospitalized
* Respiratory dysfunction defined as one Partial Arterial Oxygen Pressure to Fraction of Inspired Oxygen (PaO2/FiO2) ratio inferior to 200, independently of the Positive End Expiratory Pressure (PEEP) level.
* Total SOFA points for organ dysfunctions other than the respiratory function more than 3

Exclusion Criteria:

* Denial for informed consent
* Age inferior to 18 years
* Pregnancy (confirmed by blood or urinary pregnancy test) or lactation for female patients of reproductive age.
* Unwillingness to receive contraception during and seven days after the administration of the study drug.
* HIV infection (with known Cluster of Differentiation 4-positive [CD4] cell count ≤ 200/mm3)
* Solid organ, or bone marrow transplantation
* Corticosteroid oral or intravenous intake greater than 0.4 mg/kg of equivalent prednisone daily over the last 15 days
* Known active neoplasms compromising short-term survival (1 month)
* Neutropenia <1000/mm3
* Known allergy to macrolides
* Previous participation in the study
* Administration of a macrolide for the current infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Mortality rate at 28 days | 28 days
  Differences in early (28-day) all-cause mortality rate between clarithromycin and placebo-treated arms

SECONDARY OUTCOMES:
Mortality rate at 90 days | 90 days
  Differences in middle term (90-day) all-cause mortality rate between clarithromycin and placebo-treated arms
Mortality rate at 28 days for patients with septic shock | 28 days
  Differences in early (28-day) all-cause mortality rate between clarithromycin and placebo-treated arms in the subgroup of patients with septic shock
Rate of early sepsis response at 3 days | 3 days
  The number of patients who present at least 25% decrease of day 1 SOFA score on day 3 will be compared between clarithromycin and placebo-treated groups
Rate of sepsis resolution at 7 days | 7 days
  The number of patients who present at least 25% decrease of day 1 SOFA score on day 7 will be compared between clarithromycin and placebo-treated groups
New sepsis episode until 28 days | 28 days
  The number of patients who present a new increase of SOFA score by at least 2 points, consequent to infection, after having previously experienced sepsis resolution, will be compared between clarithromycin and placebo-treated groups
Time to new sepsis episode until 28 days | 28 days
  The time to new sepsis episode, defined as a new increase of SOFA score by at least 2 points, consequent to infection, in patients who have previously experienced sepsis resolution, will be compared between clarithromycin and placebo-treated groups
Cell population analysis | 10 days
  Flow cytometry will be compared between clarithromycin and placebo-treated arms
Transcriptome analysis | 10 days
  Expression of messenger Ribonucleic Acid (mRNA) will be compared between clarithromycin and placebo-treated arms
Metabolome analysis | 10 days
  Metabolites will be compared between clarithromycin and placebo-treated arms
Microbiome analysis | 10 days
  Gut microbiome composition will be compared between clarithromycin and placebo-treated arms
Cost of hospitalization | 28 days
  Real cost of hospitalization, i.e. medication administered and interventions performed, in euros (€), will be compared between clarithromycin and placebo-treated groups

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Armaganidis, MD, PhD, Principal Investigator — National Kapodistrian University of Athens, Medical School
Locations (12):
- Belgium (3):
  - Intensive Care Unit, Saint-Pierre University Hospital, Brussels
  - Intensive Care Unit, Brugmann University Hospital, Brussels
  - Intensive Care Unit, Erasme University Hospital, Brussels
- Greece (9):
  - Intensive Care Unit, Korgialeneio-Benakeio General Hospital, Athens
  - Intensive Care Unit, Laikon General Hospital, Athens
  - 2nd Department of Intensive Care Medicine, Attikon University Hospital, Athens
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens
  - 2nd Department of Internal Medicine, Sismanogleio General Hospital, Athens
  - Intensive Care Unit, Agios Dimitrios General Hospital, Thessaloniki
  - Intensive Care Unit, G. Gennimatas General Hospital, Thessaloniki
  - Intensive Care Unit, Theageneio Oncological Hospital, Thessaloniki
  - Intensive Care Unit, Ippokrateion General Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giamarellos-Bourboulis EJ, Mylona V, Antonopoulou A, Tsangaris I, Koutelidakis I, Marioli A, Raftogiannis M, Kopterides P, Lymberopoulou K, Mouktaroudi M, Papageorgiou C, Papaziogas B, Georgopoulou AP, Tsaganos T, Papadomichelakis E, Gogos C, Ladas M, Savva A, Pelekanou A, Baziaka F, Koutoukas P, Kanni T, Spyridaki A, Maniatis N, Pelekanos N, Kotsaki A, Vaki I, Douzinas EE, Koratzanis G, Armaganidis A. Effect of clarithromycin in patients with suspected Gram-negative sepsis: results of a randomized controlled trial. J Antimicrob Chemother. 2014 Apr;69(4):1111-8. doi: 10.1093/jac/dkt475. Epub 2013 Nov 28. PMID 24292991
- [Result] Spyridaki A, Raftogiannis M, Antonopoulou A, Tsaganos T, Routsi C, Baziaka F, Karagianni V, Mouktaroudi M, Koutoukas P, Pelekanou A, Kotanidou A, Orfanos SE, van der Meer JW, Netea MG, Giamarellos-Bourboulis EJ. Effect of clarithromycin in inflammatory markers of patients with ventilator-associated pneumonia and sepsis caused by Gram-negative bacteria: results from a randomized clinical study. Antimicrob Agents Chemother. 2012 Jul;56(7):3819-25. doi: 10.1128/AAC.05798-11. Epub 2012 May 7. PMID 22564837
- [Result] Giamarellos-Bourboulis EJ, Pechere JC, Routsi C, Plachouras D, Kollias S, Raftogiannis M, Zervakis D, Baziaka F, Koronaios A, Antonopoulou A, Markaki V, Koutoukas P, Papadomichelakis E, Tsaganos T, Armaganidis A, Koussoulas V, Kotanidou A, Roussos C, Giamarellou H. Effect of clarithromycin in patients with sepsis and ventilator-associated pneumonia. Clin Infect Dis. 2008 Apr 15;46(8):1157-64. doi: 10.1086/529439. PMID 18444850
- [Result] Tsaganos T, Raftogiannis M, Pratikaki M, Christodoulou S, Kotanidou A, Papadomichelakis E, Armaganidis A, Routsi C, Giamarellos-Bourboulis EJ. Clarithromycin Leads to Long-Term Survival and Cost Benefit in Ventilator-Associated Pneumonia and Sepsis. Antimicrob Agents Chemother. 2016 May 23;60(6):3640-6. doi: 10.1128/AAC.02974-15. Print 2016 Jun. PMID 27044546
- [Result] Schultz MJ, Speelman P, Hack CE, Buurman WA, van Deventer SJ, van Der Poll T. Intravenous infusion of erythromycin inhibits CXC chemokine production, but augments neutrophil degranulation in whole blood stimulated with Streptococcus pneumoniae. J Antimicrob Chemother. 2000 Aug;46(2):235-40. doi: 10.1093/jac/46.2.235. PMID 10933646
- [Result] Kanoh S, Rubin BK. Mechanisms of action and clinical application of macrolides as immunomodulatory medications. Clin Microbiol Rev. 2010 Jul;23(3):590-615. doi: 10.1128/CMR.00078-09. PMID 20610825
- [Derived] Karakike E, Scicluna BP, Roumpoutsou M, Mitrou I, Karampela N, Karageorgos A, Psaroulis K, Massa E, Pitsoulis A, Chaloulis P, Pappa E, Schrijver IT, Frantzeskaki F, Lada M, Dauby N, De Bels D, Floros I, Anisoglou S, Antoniadou E, Patrani M, Vlachogianni G, Mouloudi E, Antoniadou A, Grimaldi D, Roger T, Wiersinga WJ, Tsangaris I, Giamarellos-Bourboulis EJ. Effect of intravenous clarithromycin in patients with sepsis, respiratory and multiple organ dysfunction syndrome: a randomized clinical trial. Crit Care. 2022 Jun 18;26(1):183. doi: 10.1186/s13054-022-04055-4. PMID 35717241